CLINICAL TRIAL: NCT02367937
Title: A Phase I, Open-Label Study to Assess the Effects of PRC-4016 (Icosabutate) on the Pharmacokinetics of Midazolam, Omeprazole, Flurbiprofen and Simvastatin in Healthy Male/Female Subjects
Brief Title: PRC-4016 (Icosabutate) Phase I Drug-drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pronova BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CTN401614103
Record Dates: First submitted 2015-02-09; First posted 2015-02-20 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Healthy
Keywords: Phase I drug-drug interaction
MeSH Terms: interventions — icosabutate; Midazolam; Omeprazole; Flurbiprofen; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PRC-4016 (Icosabutate) (Experimental)
  Interventions: Drug: PRC-4016 (icosabutate)

INTERVENTIONS:
Drug: PRC-4016 (icosabutate) — Midazolam, omeprazole, flurbiprofen and simvastatin interaction with PRC-4016. Detailed description under "Study description"
  Other Names: Midazolam, omeprazole, flurbiprofen and simvastatin

SUMMARY:
The aim of the study is to evaluate the effect of PRC-4016 at steady state on the pharmacokinetics (PK) of cytochrome P450 (CYP) 3A substrates (midazolam, simvastatin), a CYP2C9 substrate (omeprazole) and a CYP2C19 substrate (flurbiprofen) in healthy male/female subjects.

DETAILED DESCRIPTION:
Day 1: Subject will receive single oral doses of 2.5 mg midazolam, 20 mg omeprazole and 50 mg flurbiprofen morning Day 2: Subject will receive a single oral dose of 40 mg simvastatin on the morning of Day 2. Day 4: Subjects will commence the multiple-dose regimen for PRC-4016 (600 mg once daily) for 11 days. Day 12: Subjects will be given single oral doses of 2.5 mg midazolam, 20 mg omeprazole and 50 mg flurbiprofen co-administered with 600 mg PRC-4016.

Day 13, subjects will be given a single oral dose of 40 mg simvastatin co-administered with 600 mg PRC-4016.

All subjects will return for a post-study visit 7 to 10 days after their final dose.

ELIGIBILITY:
Inclusion Criteria:

* males or females
* any ethnic origin
* age 18-60 years
* BMI 8.0 - 35.0 kg/m2
* generally good health
* signed informed consent

Exclusion Criteria:

* males or females not willing to use appropriate contraception
* recent blood donation
* recent blood received
* high consumption of alcohol
* high consumption og tobacco
* subjects who have engaged in heavy exercise last two weeks
* prescribed systemic or topical medication taken recently, or supplements/remedies interfering with study procedures or safety
* other medication known to alter drug absorption or elimination
* abnormal hearth rate or blood pressure
* significant history of drug allergy or hypersensitivity to treatment ingredients
* other significant medical history or physical findings
* pregnant or lactating
* Poor metabolizers for CYP2C9 or CYP2C19
* subjects previously taken part in or withdrawn from study or subjects that according to investigator should not participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Area under curve for effect of PRC-4016 at steady state on the PK of CYP3A substrates (midazolam, simvastatin), a CYP2C9 substrate (omeprazole) and a CYP2C19 substrate (flurbiprofen) in healthy male/female subjects. | 24 h postdose
  Blood-sampling
Peak plasma concentration for effect of PRC-4016 at steady state on the PK of CYP3A substrates (midazolam, simvastatin), a CYP2C9 substrate (omeprazole) and a CYP2C19 substrate (flurbiprofen) in healthy male/female subjects. | 24 hours post-dose
  Blood-sampling

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability of PRC-4016 co-administered with midazolam, omeprazole, flurbiprofen and simvastatin in healthy male/female subjects. | 24 h postdose
  Adverse event recording

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Chiesa, MD, Principal Investigator — Covance
Locations (1):
- Covance Clinical research Unit (CRU) Ltd,Springfield House, Hyde street, Leeds, United Kingdom